CLINICAL TRIAL: NCT01692964
Title: Clinical Evaluation of the InflammaDry Device for Detecting Dry Eye
Status: Completed | Type: Observational
Sponsor: Rapid Pathogen Screening (Industry)
Responsible Party: Sponsor
Organization: RapidPS (Unknown)
Other Study IDs: 12-0615
Record Dates: First submitted 2012-09-19; First posted 2012-09-26 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Dysfunctional Tear Syndrome
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- InflammaDry: Patients suspected of having dry eye will be tested with the InflammaDry.
  Interventions: Device: InflammaDry

INTERVENTIONS:
Device: InflammaDry — A noninvasive immunoassay for detecting MMP-9 levels in tears.

SUMMARY:
InflammaDry is a rapid diagnostic test for the detection of elevated levels of Matrix Metalloproteinase-9 (MMP-9) protein in tear fluid.

DETAILED DESCRIPTION:
The InflammaDry test will be used to aid in the diagnosis of dry eye in conjunction with other methods of clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patient voluntarily reported at least 1 episode of any of the following ocular symptoms during the last month:

  1. Burning or stinging
  2. Sandy or gritty feeling
  3. Foreign body sensation
  4. Tearing
  5. Light sensitivity
  6. Intermittent or fluctuating vision
  7. Tired eyes

Exclusion Criteria

* Allergy to cornstarch or Dacron
* Allergy to topical anesthetic or fluorescein dye
* Prior eye injury, trauma, or ocular surgery within the last 3 months
* Known blockage of the lacrimal drainage system
* Contact lens wear in the last month
* Previous corneal refractive surgery including RK, LASIK or PRK surgery
* Have an active ocular infection or history of a recent ocular infection in the last month
* Have active intraocular inflammation or history of intraocular inflammation, e.g. Uveitis
* Use of oral doxycycline, corticosteroids, or immunomodulators in the last month
* Have received topical ocular corticosteroids, topical Nonsteroidal (NSAIDs) therapy, or topical ocular cyclosporine in the last month
* Pregnant or lactating
* Use of any topical ophthalmic medications, including artificial tears 2 hours prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were clinically determined by an ophthalmic clinician to meet enrollment criteria were included in the study.
Sampling Method: Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Manatee-Sarasota Eye Clinic, Bradenton, Florida
  - Mercy Clinic - Eye Specialists, Springfield, Missouri
  - Ophthalmic Associates, Johnson City, New York
  - Ophthalmology Diagnostics & Clinical Research, El Paso, Texas

REFERENCES:
- [Derived] Sambursky R, Davitt WF 3rd, Friedberg M, Tauber S. Prospective, multicenter, clinical evaluation of point-of-care matrix metalloproteinase-9 test for confirming dry eye disease. Cornea. 2014 Aug;33(8):812-8. doi: 10.1097/ICO.0000000000000175. PMID 24977985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment took place over a 7-month period. The study was performed at private practices and academic centers.
Period: Overall Study
Arm/Group | InflammaDry
Started | 237
Completed | 237
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | InflammaDry
Number analyzed (Participants) | 237
Age, Customized [Mean (Full Range); unit: years] | 53 [18 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164
  Male | 73
Region of Enrollment [Number; unit: participants]
  United States | 237

OUTCOME MEASURES:

1. Primary Outcome: Negative and Positive Agreement of the InflammaDry at Diagnosis of Dry Eyes
Description: Negative agreement is the percentage of true negative cases compared to clinical assessment (specificity). Positive agreement is the percentage of true positive cases compared to clinical assessment (sensitivity). The InflammaDry test was compared with the clinical assessment of tear break-up time, Schirmer tear testing, and corneal staining for the confirmation of dry eye, both with and without the inclusion of the Ocular Surface Disease Index (OSDI), as a confirmatory test.
Time Frame: 20 minutes
Measure: Number (95% Confidence Interval); unit: percentage of cases
Groups:
- InflammaDry (Sensitivity): Looking for the percentage of true positives as compared to clinical assessment.
- Inflammadry (Specificity): Looking for the percentage of true negatives as compared to clinical assessment.
Arm/Group | InflammaDry (Sensitivity) | Inflammadry (Specificity)
Number analyzed (Participants) | 237 | 237
percentage of cases
  Confirmatory Testing With OSDI Inclusion | 81 [74 to 87] | 98 [91 to 100]
  Confirmatory Testing Without OSDI Inclusion | 86 [80 to 91] | 97 [91 to 99]

ADVERSE EVENTS:
Time Frame: 20 Minutes
Description: Regular monitoring by sponsor and mandatory reporting by investigator.
Arm/Group | InflammaDry
Serious Adverse Events (participants affected / at risk) | 0/237
Other Adverse Events (participants affected / at risk) | 0/237

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications shall be submitted to the Sponsor for review/comment 45 days prior to publication. Sponsor may remove confidential information. First publication shall be a multicenter study publication. Institution and/or PI may publish or present the results and data from the Institution's site individually (i) 12 months after conclusion, abandonment or termination of study at all sites, or (ii) after the Sponsor confirms there will be no multicenter study publication, whichever occurs first.